CLINICAL TRIAL: NCT05636072
Title: The WISER Study: Web Based Methods for Enhancing Resilience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00063703
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Burnout
Keywords: Burnout; Well-being; Behavioral Health
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Waitlist control group Randomized Control Design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Immediately (Experimental): Participants will engage in well-being tools immediately for 1-week.
  Interventions: Behavioral: WISER
- Waitlist Control (No Intervention): Participants will wait 1 week to begin the well-being tools.

INTERVENTIONS:
Behavioral: WISER — Participants will engage in one or more positive psychology well-being tool(s).
  Arms: Treatment Immediately

SUMMARY:
This is a research study to find out if web-based resilience tools can increase well-being.

Enrolled participants will try out one or more brief positive psychology tools. The tools ask participants to reflect on positive experiences or to do an activity (e.g., write a letter of gratitude). The study is entirely online and participants will be prompted to participate via email or text messages.

The study team is interested in the effects of the tools on stress, depression, and burnout in adults. A set of brief surveys are administered before and after using the tool, and again at follow-up periods (e.g., 1, 3, 6 and 12 months). Surveys are collected electronically using the secure, HIPAA-compliant survey software.

There is no direct benefit to participants for participating in this research study aside from the potential to experience improvements in well-being. Risks are minimal and include the potential to feel emotional or psychological distress when asked questions related to burnout.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and over are considered eligible for the study. A sub-sample will include employees (including but not limited to frontline caregivers, support staff and management) of the Duke University Health System, as well as external health systems. All participants will be invited to participate in one or more of the online tools. The investigators will allow the participation of any clinical areas/healthcare worker groups whose leaders express interest in building resilience. The investigators are targeting healthcare workers for recruitment in the study, but adults 18+ are eligible to participate in any of these tools. Identification as a healthcare worker or not is part of data collection in every tool.

Exclusion Criteria:

* Adults who are not proficient in English, do not have basic computer skills, or who have prohibitive vision or hearing disabilities will be excluded from this study as they will be incapable of full participation in the intervention and/or the survey process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Emotional Exhaustion as measured by the 5-item Emotional Exhaustion Scale | Baseline, Day 8, and 1, 6, and 12 month follow-ups
  Survey scores are measured on a 1-5 Likert-like agreement scale.

SECONDARY OUTCOMES:
Change in Emotional Recovery as measured by the 4-item Emotional Recovery Scale | Baseline, Day 8, and 1, 6, and 12 month follow-ups
  Survey scores are measured on a 1-5 Likert-like agreement scale.
Change in Work-life Integration as measured by the 7-item Work-life Integration Scale | Baseline, Day 8, and 1, 6, and 12 month follow-ups
  Survey scores are measured with a 1-4 frequency of behaviors scale.

CONTACTS AND LOCATIONS:
Overall Officials: John B Sexton, PhD, Principal Investigator — Duke
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Only the research team will be accessing the data.

REFERENCES:
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Profit J, Adair KC, Cui X, Mitchell B, Brandon D, Tawfik DS, Rigdon J, Gould JB, Lee HC, Timpson WL, McCaffrey MJ, Davis AS, Pammi M, Matthews M, Stark AR, Papile LA, Thomas E, Cotten M, Khan A, Sexton JB. Randomized controlled trial of the "WISER" intervention to reduce healthcare worker burnout. J Perinatol. 2021 Sep;41(9):2225-2234. doi: 10.1038/s41372-021-01100-y. Epub 2021 Aug 9. PMID 34366432
- [Background] Adair KC, Kennedy LA, Sexton JB. Three Good Tools: Positively reflecting backwards and forwards is associated with robust improvements in well-being across three distinct interventions. J Posit Psychol. 2020;15(5):613-622. doi: 10.1080/17439760.2020.1789707. Epub 2020 Jul 9. PMID 34295357
- [Background] Sexton JB, Adair KC, Cui X, Tawfik DS, Profit J. Effectiveness of a bite-sized web-based intervention to improve healthcare worker wellbeing: A randomized clinical trial of WISER. Front Public Health. 2022 Dec 8;10:1016407. doi: 10.3389/fpubh.2022.1016407. eCollection 2022. PMID 36568789
- [Background] Sexton JB, Adair KC. Well-Being Outcomes of Health Care Workers After a 5-Hour Continuing Education Intervention: The WELL-B Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2434362. doi: 10.1001/jamanetworkopen.2024.34362. PMID 39298170